CLINICAL TRIAL: NCT00537550
Title: GIMEMA Guidelines for the Treatment of Adult ALL Affected Patients at Diagnosis
Brief Title: Adult ALL Treatment at Diagnosis
Acronym: LAL2000
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LAL2000
Record Dates: First submitted 2007-09-27; First posted 2007-10-01 (Estimated); Last update posted 2007-10-01 (Estimated); Status verified 2007-09

CONDITIONS: Leukemia, Lymphocytic, Acute
Keywords: ALL; Adult
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Vincristine; Daunorubicin; Asparaginase; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Vincristine — Steroids pre-treatment
Drug: Vincristin, Daunorubicine, Asparaginase, Methotrexate — Induction therapy

SUMMARY:
The present study has been designed to give participating centers the possibility of better understanding the diagnostic and prognostic factors of ALL patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute lymphoblastic leukemia (ALL)
* Negative myeloperoxidase stain
* Phenotype T (ALL-T) and B(ALL-B)

Exclusion Criteria:

* Creatinine > 2.5mg/dL after adequate hydratation
* LVEF <50%
* Presence of documented infections not responding to antibiotic and/or antifungal therapy
* Presence of concomitant malignant diseases
* Absence of any psychological condition that does not allow to intake high doses of cortisone
* Patients who have received any antineoplastic chemiotherapy for more than 5 days
* Patients who have received any steroids for more than 10 days

Ages: 14 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 2000-07; Study Completion 2006-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Franco MANDELLI, Pr, Principal Investigator — Università degli Studi di Roma "La Sapienza"
Locations (5):
- Italy (5):
  - Az. Ospedaliera S. G. Moscati, Avellino
  - Ist.Ematologia e Oncologia Medica L.e A. Seragnoli, Bologna
  - Ospedale Reg. A di Summa, Brindisi
  - Istituto di Ematologia- Ospedale San Carlo, Potenza
  - Policlinico G.B. Rossi, Verona

REFERENCES:
- [Derived] Piciocchi A, Messina M, Elia L, Vitale A, Soddu S, Testi AM, Chiaretti S, Mancini M, Albano F, Spadano A, Krampera M, Bonifacio M, Cairoli R, Vetro C, Colella F, Ferrara F, Cimino G, Bassan R, Fazi P, Vignetti M. Prognostic impact of KMT2A-AFF1-positivity in 926 BCR-ABL1-negative B-lineage acute lymphoblastic leukemia patients treated in GIMEMA clinical trials since 1996. Am J Hematol. 2021 Sep 1;96(9):E334-E338. doi: 10.1002/ajh.26253. Epub 2021 Jun 9. No abstract available. PMID 34048072